CLINICAL TRIAL: NCT04785742
Title: An Open, Multicenter Phase II Clinical Study to Evaluate the Safety and Efficacy of Almonertinib in Patients With Advanced NSCLC With Rare Mutations in EGFR
Brief Title: Almonertinib for Advanced NSCLC Patients With Rare Mutations in EGFR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Chief Physician, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: YX-L-202008
Record Dates: First submitted 2021-01-25; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Safety of Almonertinib
MeSH Terms: interventions — aumolertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20 exon (20INS) mutation (Experimental)
  Interventions: Drug: Almonertinib
- Rare mutations except for 20INS (Experimental)
  Interventions: Drug: Almonertinib

INTERVENTIONS:
Drug: Almonertinib — Almonertinib

SUMMARY:
This is a multicenter, open, phase II clinical trial evaluating the safety and efficacy of high-dose almonertinib in the treatment of rare mutations in locally advanced or metastatic NSCLC patients with EGFR mutations (excluding exon 19 deletion or rare mutations outside L858R). Patients showed EGFR mutations by tissue or blood tests (excluding exon 19 deletion or rare mutations other than L858R), of which 20 exon (20INS) mutations and rare mutations other than 20Ins were classified as two covariates. High-dose amitinib was used for treatment to evaluate the safety and efficacy of the treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 ≤ age ≤75, regardless of gender. 2. Histologically confirmed locally advanced or metastatic non-scaly NSCLC (including stage IIIB-IV patients who relapsed after previous surgical treatment or were newly diagnosed). According to AJCC edition 8 lung cancer staging criteria).

  3. Previous treatment with second-line chemotherapy (no EGFR-TKI) is allowed. 4. Positive EGFR driver mutation (rare mutation other than 19 exon deletion or L858R) detected by tumor tissue or blood samples.

  5. The Eastern Tumor Tissue Cooperative Group (ECOG) physical status score was 0 or 1 and did not deteriorate in the previous 2 weeks, with a minimum expected survival of 12 weeks.

  6. The patient had at least one tumor lesion that had not received previous local treatment such as irradiation, nor had he received biopsy during the screening period, and it could be accurately measured at baseline, with the longest diameter ≥ 10mm at baseline (short diameter ≥ 15mm for lymph nodes). The measurement method chosen is suitable for accurate repeated measurements and can be computed tomography (CT) or magnetic resonance imaging (MRI). If there is only one measurable lesion and no previous local treatment such as irradiation, it may be accepted as the target lesion, and a baseline evaluation of the tumor lesion shall be conducted at least 14 days after the diagnostic biopsy.

  7. For fertile women, appropriate contraception should be used and breastfeeding should not be performed for 3 months from screening to discontinuation of study treatment. A pregnancy test is negative before administration, or there is no proven risk of pregnancy if one of the following criteria is met:

A. Postmenopause is defined as amenorrhea over the age of 50 and at least 12 months after cessation of all exogenous hormone replacement therapy.

B. Women younger than 50 years of age may also be considered postmenopausal if they stop all exogenous hormone therapy for 12 months or more and their luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels are within the laboratory post-menopausal reference range.

C. Has undergone irreversible sterilization, including hysterectomy, bilateral oophorectomy or bilateral salpingectomy, except for bilateral tubal ligation.

8. Male patients should use barrier contraception (i.e., condoms) from screening until 3 months after treatment is discontinued.

9. The subject is willing to participate and sign the informed consent in person.

Exclusion Criteria:

* 1. Have received any of the following treatments:

A. Patients who underwent major surgery within 4 weeks prior to the first dosing of the study drug;

B. Patients who received more than 30% bone marrow irradiation or received large area radiotherapy within 4 weeks prior to the first dosing of the study drug;

C. Study drugs that had used a CYP3A4 inhibitor, inducer, or a narrow therapeutic window with a CYP3A4-sensitive substrate within 7 days before first administration.

2. Patients with other malignancies requiring standard treatment or major surgery within 2 years of the first dosing of study therapy.

3. At the start of the study, there were unmitigated residual toxicity from previous treatment greater than CTCAE grade 1, except for grade 2 neurotoxicity caused by hair loss and previous chemotherapy.

4. Spinal cord compression or brain metastasis, unless asymptomatic, stable, and does not require steroid therapy for at least 2 weeks prior to first dosing of study therapy.

5. Any serious or poorly controlled systemic disease, as determined by the investigator, such as poorly controlled hypertension, active bleeding susceptibility, or active infection. There is no need to screen for chronic diseases.

6. Full absorption of amitinib may be affected by refractory nausea, vomiting, or chronic gastrointestinal disorders, inability to swallow study drugs, or previous extensive enterectomy.

7. Satisfy one of the following cardiac test results:

A. Average corrected QT interval (QTC) > 470 msec from three resting electrocardiogram (ECG) examinations, QT interval correction (QTCF) was performed using Fridericia's formula;

B. Resting ECG suggests the presence of a variety of clinically significant rhythm, conduction, or ECG morphological abnormalities (such as complete left bundle branch block, degree 3 atrioventricular block, degree 2 atrioventricular block, and PR interphase > 250 Msec);

C. The presence of any factors that increase the risk of prolonged QTC or arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, a family history of long QT syndrome or sudden unexplained death of an immediate family member under 40 years of age, or any combination drug that prolongs QT interval;

D. Left ventricular ejection fraction (LVEF) ≤40%.

8. Any history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonia requiring steroid treatment, or evidence of clinically active interstitial lung disease.

9. Bone marrow reserve or organ function is insufficient, reaching the following laboratory limits:

A. Hypoalbuminemia:Absolute neutrophil count <1.5×109 / L;

B. Thrombocytopenia:Platelet count <100×109 / L;

C. Hypoproteinemia:Hemoglobin <90 g/L (<9 g/dL);

D.Liver dysfunction.If there is no definite liver metastasis, alanine aminotransferase > is 2.5 times the upper normal limit (ULN); If there is liver metastasis, alanine aminotransferase > 5×ULN;

E. Liver dysfunction.If there is no definite liver metastasis, aspartic aminotransferase > 2.5×ULN; If there is liver metastasis, aspartate aminotransaminase > 5×ULN.

F. Hyperbilirubinemia.If there is no definite liver metastasis, total bilirubin > 1.5×ULN; Or Gilbert syndrome (unbound hyperbilirubinemia) or liver metastasis, total bilirubin > 3×ULN;

G. Creatinine > 1.5×ULN and creatinine clearance <50 mL/min (calculated by Cockcroft - Gault formula); Creatinine clearance needs to be confirmed only when creatinine > 1.5×ULN.

10. Women who are lactating or who have positive blood or urine pregnancy test results within 3 days prior to the first dosing of study treatment.

11.Hypersensitivity: A history of hypersensitivity to any active or inactive ingredient of almonertinib or to drugs similar in chemical structure to or similar to almonertinib.

12. Any serious or uncontrolled ocular lesions that may, in the judgment of the physician, increase the patient's safety risk.

13. Patients identified by the investigator as likely to have poor compliance with study procedures and requirements.

14. Patients identified by the investigator as having any condition that jeopardizes patient safety or interferes with study evaluation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 36 months
  To evaluate the security of high-dose Almonertinib for advanced NSCLC patients with rare mutations in EGFR

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No